CLINICAL TRIAL: NCT03039803
Title: Impact of Double-layer Versus Single-layer Uterine Closure Suture in Cesarean Section on the Development of Postoperative Uterine Scar Deficiency: A Randomized Controlled Trial
Brief Title: Impact of Double-layer Versus Single-layer Uterine Closure Suture in Cesarean Section on the Development of Postoperative Uterine Scar Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Samir Helmy, Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1642/2016
Record Dates: First submitted 2016-11-27; First posted 2017-02-01 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Cesarean Section; Uterine Scar Deficiency; Myometrial Thickness; Single-layer Continuous Uterotomy Suture; Double-layer Continuous Uterotomy Suture; Transvaginal Ultrasound

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- single-layer continuous uterotomy suture (Active Comparator): Single-layer continuous uterotomy suture
  Interventions: Procedure: uterine closure during cesarean section
- double-layer continuous uterotomy suture (Active Comparator): double-layer continuous uterotomy suture
  Interventions: Procedure: uterine closure during cesarean section

INTERVENTIONS:
Procedure: uterine closure during cesarean section

SUMMARY:
In recent decades, the rate of cesarean section delivery has steadily increased worldwide ranging at 30% of deliveries, thus long-term risks after cesarean section need to be evaluated. Postoperative risks include, among others, uterine scar rupture and placental complications such as placenta previa and accreta- complications, which are possibly associated with uterine scar dehiscence.

The prevalence of lower-segment uterine scar deficiency has previously been described as 63%. One recent systematic review and meta analysis investigated closure techniques of low transverse cesarean. No significant difference in risk of uterine scar defect comparing single layer versus double layer closure could be detected (RR 0.53), whereas in women with single layer closure, a lower residual myo-metrial thickness was observed (-2.6mm). However, the authors do conclude that data is insufficient to determine the risk of uterine rupture, dehiscence or gynecological outcomes due to insufficient power of available studies. A recently published Randomized Controlled Trial concluded that double-layer closure with unlocked first layer showed a better scar healing than locked single layer.

The investigators main objective is to identify if single-layer suture of the uterus during cesarean section results in a higher rate of cesarean scar deficiency than double-layer suture.

Interventions

Single- layer versus double- layer uterine closure Two different techniques of uterine closure in cesarean section will be compared: single- layer versus double- layer continuous uterotomy suture.

Standardized transvaginal sonography

Transvaginal ultrasound examination is carried out by one expert sonographer. The ultrasound machine used for all examinations is GE Voluson E10.

Primary outcome: CS scar deficiency visualized in transvaginal ultrasound at 3 months after CS (yes/no).

Secondary outcome: Myometrial thickness at the site of uterine scar (mm).

ELIGIBILITY:
Inclusion Criteria:

* First cesarean section
* Scheduled cesarean section at Department of Obstetrics and Gynecology, Medical University of Vienna
* Age ≥ 18 years
* Informed Consent
* Cesarean section at ≥ 37+0 weeks of gestation

Exclusion Criteria:

* Previous cesarean section
* Emergency cesarean section
* Cesarean section < 37+0 weeks of gestation
* Corporal incision during cesarean section
* Diseases which favor wound healing disruptions (e.g. chronic inflammatory diseases)
* Uterine anatomic anomalies
* BMI > 35kg/m2
* Placenta previa

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Cesarean section (CS) scar deficiency visualized in transvaginal ultrasound at 3 months after CS (yes/no). | 3 months

SECONDARY OUTCOMES:
Myometrial thickness at the site of uterine scar (mm). | 3 months

OTHER OUTCOMES:
The presence or absence of a CS scar pregnancy in a consecutive pregnancy | up to 25 years
Occurence of uterine rupture in a consecutive pregnancy | up to 25 years
CS scar deficiency visualized in transvaginal ultrasound (yes/no) in early pregnancy in a consecutive pregnancy | up to 25 years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Ofili-Yebovi D, Ben-Nagi J, Sawyer E, Yazbek J, Lee C, Gonzalez J, Jurkovic D. Deficient lower-segment Cesarean section scars: prevalence and risk factors. Ultrasound Obstet Gynecol. 2008 Jan;31(1):72-7. doi: 10.1002/uog.5200. PMID 18061960
- [Background] Roberge S, Demers S, Berghella V, Chaillet N, Moore L, Bujold E. Impact of single- vs double-layer closure on adverse outcomes and uterine scar defect: a systematic review and metaanalysis. Am J Obstet Gynecol. 2014 Nov;211(5):453-60. doi: 10.1016/j.ajog.2014.06.014. Epub 2014 Jun 6. PMID 24912096
- [Background] Clark SL, Koonings PP, Phelan JP. Placenta previa/accreta and prior cesarean section. Obstet Gynecol. 1985 Jul;66(1):89-92. PMID 4011075
- [Background] Gilliam M, Rosenberg D, Davis F. The likelihood of placenta previa with greater number of cesarean deliveries and higher parity. Obstet Gynecol. 2002 Jun;99(6):976-80. doi: 10.1016/s0029-7844(02)02002-1. PMID 12052584
- [Background] Miller DA, Chollet JA, Goodwin TM. Clinical risk factors for placenta previa-placenta accreta. Am J Obstet Gynecol. 1997 Jul;177(1):210-4. doi: 10.1016/s0002-9378(97)70463-0. PMID 9240608
- [Background] Silver RM. Abnormal Placentation: Placenta Previa, Vasa Previa, and Placenta Accreta. Obstet Gynecol. 2015 Sep;126(3):654-668. doi: 10.1097/AOG.0000000000001005. PMID 26244528
- [Background] Thurn L, Lindqvist PG, Jakobsson M, Colmorn LB, Klungsoyr K, Bjarnadottir RI, Tapper AM, Bordahl PE, Gottvall K, Petersen KB, Krebs L, Gissler M, Langhoff-Roos J, Kallen K. Abnormally invasive placenta-prevalence, risk factors and antenatal suspicion: results from a large population-based pregnancy cohort study in the Nordic countries. BJOG. 2016 Jul;123(8):1348-55. doi: 10.1111/1471-0528.13547. Epub 2015 Jul 29. PMID 26227006
- [Background] Roberge S, Demers S, Girard M, Vikhareva O, Markey S, Chaillet N, Moore L, Paris G, Bujold E. Impact of uterine closure on residual myometrial thickness after cesarean: a randomized controlled trial. Am J Obstet Gynecol. 2016 Apr;214(4):507.e1-507.e6. doi: 10.1016/j.ajog.2015.10.916. Epub 2015 Nov 11. PMID 26522861
- [Background] Dodd JM, Anderson ER, Gates S, Grivell RM. Surgical techniques for uterine incision and uterine closure at the time of caesarean section. Cochrane Database Syst Rev. 2014 Jul 22;2014(7):CD004732. doi: 10.1002/14651858.CD004732.pub3. PMID 25048608